CLINICAL TRIAL: NCT03122080
Title: Efficacy and Safety of Electroacupuncture on Treating Depression Related Insomnia: Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Efficacy of EA on Depression Related Insomnia: Study Protocol for a Multicenter RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other); Changhai Hospital (Other); Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHMHTCM Shifen Xu
Record Dates: First submitted 2017-03-20; First posted 2017-04-20 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Insomnia Due to Mental Disorder
Keywords: acupuncture; insomnia; depression; antidepressants
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Electroacupuncture; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture group (Active Comparator): electroacupuncture+standard care
  Interventions: Device: Electroacupuncture(EA)
- Control A group (Placebo Comparator): placebo acupuncture+standard care
  Interventions: Device: Placebo acupuncture
- Control B group (Other): standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Electroacupuncture(EA) — Participants in EA group will receive electroacupuncture treatment. Acupuncture will be applied at Baihui (GV20), Shenting (GV24), Yintang (GV29), bilateral Anmian (EX-HN22), Shenmen (HT7), SanYinjiao (SP6) and Neiguan (PC6). After needle insertion, rotating or lifting-thrusting manipulation will be applied for "Deqi" sensation. The EA apparatus (CMNS6-1, Jianjian Medical Device CO., LTD, China) will be connected to the needles at GV20 and GV29 for 30 minutes and deliver a continuous wave. The frequency will be set at about 30 Hz and the amplitude will be less than 20V. Participants can regularly take the antidepressants or sedative-hypnotics as before during the intervention. Besides, the investigators will strengthen health education about insomnia and depression for the patients.
  Arms: Electroacupuncture group
Device: Placebo acupuncture — Participants in the control A group will receive placebo acupuncture treatment with streitberger needles at the same acupoints as the electroacupuncture group. When the tip of the blunt needles touches to the skin, the patient will get a pricking sensation but there is no real needle inserted into the skin. The electroacupuncture apparatus will be set beside the patients, with no connection to the needles. Inform the patients when removing the needles after 30 minutes. Use the dry cotton ball to press the acupoints so that patients can feel the withdrawal of the 'needles'. Same health education and regular administration of antidepressants or sedative-hypnotics will be given to the participants during the intervention.
  Arms: Control A group
Other: Standard care — Participants in the control B group will keep their standard medical care for the first 8 weeks. Participants will take their regular antidepressants and the sedative-hypnotics during the whole intervention period. Same health education will be conducted as well for the participants. And after waiting for two months, these patients will be treated with the same electroacupuncture treatment as the EA group.
  Arms: Control B group

SUMMARY:
The investigators describe a protocol for a multicenter randomized controlled trial to find out the efficacy of electroacupuncture for depression related insomnia.

DETAILED DESCRIPTION:
Sleep difficulties are among the main symptoms presented by depressed patients, and they can profoundly impact course of illness. Acupuncture is a widely recognized therapy to treat depressive disorders and sleep disturbances in clinical practice. This multicenter randomized placebo-controlled trial is aimed to investigate the efficacy and safety of electroacupuncture, sham acupuncture and standard medical care, administrated by professional acupuncturists and psychiatrists, in depression patients with insomnia.

The investigators describe a protocol for a multicenter randomized controlled trial. Two hundred seventy eligible patients in 3 different health-care centers in Shanghai will be randomly assigned to one of 3 treatment groups: EA group (electroacupuncture+standard medical care), Control A group (sham acupuncture+standard medical care) and Control B group (standard medical care). Treatment will be given 3 times per week for 8 weeks. The primary outcomes is the Pittsburgh Sleep Quality Index (PSQI). The secondary outcomes are sleep parameters recorded in the Actigraphy, Hamilton Rating Scale for Depression (HAMD) score and Self-rating Anxiety Scale (SAS) score. Daily dose of patients' antidepressant and sedative-hypnotic medication will be recorded in the dairy. All adverse effects will be assessed by the Treatment Emergent Symptom Scale (TESS). Outcomes will be evaluated at baseline, 4 weeks post-treatment and 8 weeks post-treatment, as well as at 1 month, 3 months and 6 months follow-up.

The findings from this trial will help further about the efficacy and safety of acupuncture for depression related insomnia, as well as determine the differences between electroacupuncture, sham acupuncture and standard medical care for treating insomnia and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18-70;
2. Participants who meet the diagnostic criteria of depression according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV);
3. Participants whose HAMD score is 20-35;
4. Participants who have complaint about insomnia at the first visit to the doctor;
5. Participants whose PSQI score is more than 7;
6. Participants who voluntarily agree with the investigation and sign a written informed consent form for the clinical trial.

Exclusion Criteria:

1. Participants with secondary depressive disorders caused by organic diseases, medicine, or psychotic disorders including schizophrenia, etc;
2. Participants who are in the depressive episode of bipolar disorder, or suffering from dysthymia, reactive depression and depressive syndrome caused by other diseases;
3. Participants with alcohol abuse or drug dependence;
4. Participants who refuse to wear the Actigraphy during the trial;
5. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 8 week post-treatment
  The Pittsburgh Sleep Quality Index (PSQI) is a widely-used questionnaire to assess one's sleep disorders over one month. It is comprised of 19 self-rated items and 5 other-rated items. The scores include the following indicators: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of medication, and daytime dysfunction. Each indicator is rated from 0 to 3. The accumulated scores of the seven indicators constitute the total score of PSQI (0-21). The higher score indicates the worse sleep quality and severer sleep disorders. The investigators set the PSQI score at 8th week post-treatment as the primary outcome, compared with PSQI scores at other time points, to evaluate the effectiveness of acupuncture for depression related insomnia.

SECONDARY OUTCOMES:
Changes of PSQI scores from baseline to 6 month follow-up | baseline, 4 week post-treatment, 8 week post-treatment, 1 month,3 month, 6 month follow-up
  As is mentioned above, PSQI is a widely-used questionnaire to assess one's sleep disorders over one month. In order to assess the effects of acupuncture on patients' sleep quality during the intervention period, and to assess the durative effects of acupuncture after the intervention ends, the investigators set the changes of PSQI scores between baseline to 6 month follow-up as the secondary outcome.
Actigraphy | baseline, 4 week post-treatment, 8 week post-treatment
  Actigraphy (wActiSleep-BT. LLC, Pensacola, USA), which is worn on the patient's wrist, can monitor the quality of sleep, such as sleep onset, sleep latency, total sleep time, sleep awakenings during the night, duration of sleep, and sleep efficiency. The software ActiLife6 (Version 6.8.1, ActiGraph, LLC) will be used to analyze every participant's sleep condition recorded in the actigraphy.
Hamilton Rating Scale for Depression (HAMD) | baseline, 4 week post-treatment, 8 week post-treatment, 1 month, 3 month, 6 month follow-up
  The Hamilton Rating Scale for Depression (HAMD), an observer-rating questionnaire with 17 items to describe the severity of cognitive and bodily symptoms of depressive disorders. Each item is rated in 3- or 5-point scales. The higher total score indicates the severer depression.
Self-rating Anxiety Scale (SAS) | baseline, 4 week, 8 week post-treatment
  The Self-rating Anxiety Scale (SAS) is primarily used as a measure of somatic symptoms associated with anxiety. In using the scale, the participant will be asked to rate each item from 0-3 points according to how it applies to him or her within the past week. The standard score is the sum of the integer part of 1.25 times the raw score of the 20 items. A standard score of more than 50 points means the subject has anxious symptoms. A higher score indicates a more serious case of anxiety.
Dose dairy | baseline, 4 week, 8 week post-treatment, 1 month, 3 month, 6 month follow-up
  The dose dairy is a notebook where participants will be required to record their daily dose of antidepressants or sedative-hypnotics from baseline to 6 months follow-up, as well as the dosage time.

OTHER OUTCOMES:
Adverse effects | baseline, 4 week post-treatment, 8 week post-treatment, 1 month, 3 month, 6 month follow-up.
  Any adverse event (described as unfavourable or unintended signs, symptoms or diseases occurring during the trial) related to the intervention or administration of antidepressants and sedative-hypnotics will be reported by patients and practitioners and accessed by the Treatment Emergent Symptom Scale (TESS) which is used as an associated indicator to mainly evaluate the safety of acupuncture treatment in this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shifen Xu, PhD, Study Director — Shanghai Municipal Hospital of TCM; Xia Li, Principal Investigator — Shanghai Mental Health Center; Shuang Zhou, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yin X, Li W, Liang T, Lu B, Yue H, Li S, Zhong VW, Zhang W, Li X, Zhou S, Mi Y, Wu H, Xu S. Effect of Electroacupuncture on Insomnia in Patients With Depression: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220563. doi: 10.1001/jamanetworkopen.2022.20563. PMID 35797047
- [Derived] Yin X, Dong B, Liang T, Yin P, Li X, Lin X, Zhou S, Qian X, Lao L, Xu S. Efficacy and safety of electroacupuncture on treating depression-related insomnia: a study protocol for a multicentre randomised controlled trial. BMJ Open. 2019 Apr 20;9(4):e021484. doi: 10.1136/bmjopen-2018-021484. PMID 31005904